CLINICAL TRIAL: NCT02883361
Title: Motivational Enhancement Therapy to Improve Adherence to Aromatase Inhibitors
Acronym: MI for AIs
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Our team decided to conduct more preliminary work on understanding AI adherence to support the optimal development of a randomized controlled trial before proceeding with the trial.
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB16-1463
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Medication Adherence
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Receive 4 in-person motivational enhancement counseling sessions over the course of 12-months that specifically target medication adherence.
  Interventions: Behavioral: Motivational enhancement therapy
- Control (Placebo Comparator): Attend 4 in-person sessions to complete questionnaires and receive educational handouts.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Motivational enhancement therapy — Counseling meant to enhance motivation and decrease ambivalence about change, including asking open-ended questions, eliciting change-talk, and identifying discrepancies between current behaviour and valued behaviour
  Other Names: Motivational interviewing
  Arms: Treatment
Behavioral: Attention Control — Having participants come into the lab and fill out questionnaires with a researcher in-person
  Arms: Control

SUMMARY:
The proposed research is a randomized controlled investigation of the efficacy of motivational interviewing (MI) to improve adherence to aromatase inhibitors (AI) in a community sample of patients with poor adherence to AIs.

DETAILED DESCRIPTION:
Background: The use of Aromatase Inhibitors (AIs) among breast cancer (BC) patients with hormone receptor-positive disease reduces recurrence by 41% and mortality by 31%. Despite the efficacy of AIs, one-quarter of BC survivors fail to take their AIs as prescribed during the first year with another one-fifth discontinuing later in treatment. There are a variety of reasons for non-adherence, including low motivation, poor patient-provider communication, low self-efficacy, low perceived risk, and the experience of side effects. One promising intervention for improving treatment adherence is motivational interviewing (MI), a broad set of patient-centered techniques designed to enhance motivation for behaviour change. Objectives: To conduct a parallel-group, double-blind, randomized controlled trial (RCT) to evaluate the efficacy of MI at improving 12-month adherence to AIs relative to attention control (AC). The primary outcome is medication adherence measured using pharmacy records and calculated by medication possession ratio (MPR). Secondary outcomes include self-reported adherence, motivation and self-efficacy. Methods: A community sample of BC survivors newly prescribed AIs will be recruited from a local cancer centre pharmacy for a 6-month medication adherence observation period. The investigators chose to recruit new AI users because a significant number (i.e., 20-35%) are expected to discontinue medication within 12-months. MPR will be calculated following the observation period and patients meeting inclusion criteria and deemed non-adherent (MPR < 80%) will be enrolled in the trial, randomly assigned to MI or AC, and scheduled for a baseline appointment. Recruitment will continue until 128 (64 per group) non-adherent BC survivors are identified. Four MI or AC sessions will be delivered at 3-month intervals (0-,3-,6-,9-months), each lasting 30-45 minutes. A final assessment will occur at 12-months. Baseline and final assessments will be conducted by an assistant who is not affiliated with the trial. Given that the long-term adherence to AIs is poor, a lack of adherence leads to clinically meaningful increases in BC recurrence, morbidity and mortality, and there has been only one published intervention study related to AIs to date, our trial represents a top priority in the prevention and treatment of BC.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women, prescribed their first aromatase inhibitor medication. Been identified as non-adherent following a 6-month observation run-in period (Phase 1).

Exclusion Criteria:

* Unable to comply with protocols; diagnosis of cognitive impairment; severe psychopathology (e.g., schizophrenia); history of drug abuse; terminal condition with low likelihood of survival; living in a long-term care facility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence measured using medication possession ratio (MPR) | 12-months

SECONDARY OUTCOMES:
Motivation for medication adherence | 12-months
  Change in motivation measured using the Treatment Self Regulation Questionnaire
Self-report medication adherence | 12-months
  Change in self-report medication adherence

OTHER OUTCOMES:
Self Efficacy for Medication Adherence | 12-months
  Change in self-efficacy for medication adherence measured using the Medication Adherence Self Efficacy Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural Medicine Laboratory, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided